CLINICAL TRIAL: NCT07295158
Title: Laparoscopic Cholecystectomy Patients: Effect of Sevoflurane vs. Desflurane on Mechanical Power - A Prospective, Randomized, Controlled Trial
Brief Title: Effect of Sevoflurane vs Desflurane on Mechanical Power in Laparoscopic Cholecystectomy
Acronym: VAPOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Nuran Akıncı Ekinci, Specialist in Anesthesiology and Reanimation, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LC-MP-2025-01"
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Perioperative Respiratory Mechanics
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and postoperative outcome assessors are masked to group allocation. The anesthesia team administering sevoflurane or desflurane is not blinded, but all intraoperative data collectors and postoperative evaluators remain blinded to the inhalational agent used. Randomization is performed using sealed opaque envelopes to maintain allocation concealment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm S- Sevoflurane Group (Experimental): Maintenance of general anesthesia with sevoflurane 2% during laparoscopic cholecystectomy. Mechanical power is measured at three intraoperative time points using standardized ventilator settings.
  Interventions: Drug: Sevoflurane
- Arm D-desflurane group (Experimental): Maintenance of general anesthesia with desflurane 6% during laparoscopic cholecystectomy. Mechanical power is measured at three standardized intraoperative time points under identical ventilator settings.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — General anesthesia will be maintained with sevoflurane at 2% concentration in patients assigned to the Sevoflurane Group (Group S). Standardized ventilator settings will be applied for all participants, and mechanical power will be measured at three intraoperative time points while sevoflurane is used as the sole maintenance inhalational agent.
  Other Names: Group S
  Arms: Arm S- Sevoflurane Group
Drug: Desflurane — Maintenance of general anesthesia with desflurane 6% during laparoscopic cholecystectomy. Mechanical power is measured at three intraoperative time points using standardized ventilator settings.
  Arms: Arm D-desflurane group

SUMMARY:
This single-center, prospective, randomized, assessor-blinded clinical trial aims to compare the effects of sevoflurane and desflurane anesthesia on intraoperative mechanical power in adult patients undergoing elective laparoscopic cholecystectomy. Mechanical power will be measured at three standardized time points using a validated formula, and secondary outcomes include driving pressure values and early postoperative respiratory complications (desaturation, laryngospasm, bronchospasm, cough).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years

ASA Physical Status I-II

Scheduled for elective laparoscopic cholecystectomy

Able to provide written informed consent

Exclusion Criteria:

Known hypersensitivity or contraindication to study medications (sevoflurane or desflurane)

Severe chronic obstructive pulmonary disease (COPD)

Uncontrolled bronchial asthma

Decompensated heart failure (NYHA Class III-IV)

History of prior lung surgery

Morbid obesity (BMI > 35 kg/m²)

Pregnancy

Refusal to participate or inability to provide informed consent

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Mechanical Power (MP) during General Anesthesia | Measured at three intraoperative time points: Post-intubation baseline (MP1) 15 minutes after pneumoperitoneum (MP2) End of surgery before emergence (MP3)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jo YY, Chang YJ, Lee D, Kim YB, Jung J, Kwak HJ. Comparisons of Mechanical Power and Respiratory Mechanics in Pressure-Controlled Ventilation and Volume-Controlled Ventilation during Laparoscopic Cholecystectomy in Elderly Patients. J Pers Med. 2023 Jan 23;13(2):201. doi: 10.3390/jpm13020201. PMID 36836435